CLINICAL TRIAL: NCT02838056
Title: Early Detection of the Effect of Epidural Local Anesthetic by Temperature Change on the Big Toe
Brief Title: Early Detection of Epidural Onset by Temperature Change
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 201505007
Record Dates: First submitted 2016-07-12; First posted 2016-07-20 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2016-05

CONDITIONS: Early Confirmation of Epidural Catheterization
Keywords: anesthesia, epidural; skin temperature
MeSH Terms: interventions — Injections, Epidural

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- epidural injection (Experimental): epidural injection of 2% lidocaine 17 ml + 2 ml alfentanil (544 mcg x 2 = 1088 mcg) + 7% sodium bicarbonate 2.3 ml (1.9 mEq) + 0.1mg epinephrine (1:200000)
  Interventions: Drug: epidural injection

INTERVENTIONS:
Drug: epidural injection — drug combination: 2% lidocaine 17 ml + 2 ml alfentanil (544 mcg x 2 = 1088 mcg) + 7% sodium bicarbonate 2.3 ml (1.9 mEq) + 0.1mg epinephrine (1:200000)

SUMMARY:
Traditionally, placement of the epidural catheter is based on hand feel of passing through the ligamentum flavum as well as "loss of resistance" while injecting the air through the needle. However, both are subjective and not necessarily encountered consistently. Moreover, the onset of sensory block is usually slow, thus making confirmation of catheter position a tough task and may delay the turnover of the operating room. The only way to confirm the catheter position objectively without delaying surgery is to find a reliable indicator within minutes of local anesthetic injection. In this study, we try to use the change of temperature in the big toe as a surrogate indicator of correct epidural catheterization.

DETAILED DESCRIPTION:
Epidural anesthesia loading dose: 17ml 2% xylocaine + 2.3ml sodium bicarbonate + 2ml Rapifen (1088 mcg) + 0.1 mg epinephrine

ELIGIBILITY:
Inclusion Criteria:

* Body weight:50-90kg,
* American Society of Anesthesiologists physical status classification I-II,
* Under epidural anesthesia for surgery

Exclusion Criteria:

* History of receiving lumbar surgery
* Allergy to alfentanil ,xylocaine, bicarbonate
* Trauma

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-02-21 (Actual); Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
measurement of skin temperature change over big toe after epidural local anesthetic injection | within 10 mins after injection
  SPECTRUM 9000MB to detect lower limb color changes

SECONDARY OUTCOMES:
measurement of skin sensation change between inguinal area to umbilicus | within 15 mins after injection
  tested by alcohol sponge

CONTACTS AND LOCATIONS:
Overall Officials: Jui-An Lin, MD, Principal Investigator — Taipei Medical University/Wan Fang Hospital
Locations (1):
- Taipei Medical University/Wan Fang Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cherng CH, Wong CS, Ho ST. Epidural fentanyl speeds the onset of sensory block during epidural lidocaine anesthesia. Reg Anesth Pain Med. 2001 Nov-Dec;26(6):523-6. doi: 10.1053/rapm.2001.27852. PMID 11707790
- [Background] Werdehausen R, Braun S, Hermanns H, Freynhagen R, Lipfert P, Stevens MF. Uniform distribution of skin-temperature increase after different regional-anesthesia techniques of the lower extremity. Reg Anesth Pain Med. 2007 Jan-Feb;32(1):73-8. doi: 10.1016/j.rapm.2006.07.009. PMID 17196496
- [Background] Coda BA, Brown MC, Schaffer R, Donaldson G, Jacobson R, Hautman B, Shen DD. Pharmacology of epidural fentanyl, alfentanil, and sufentanil in volunteers. Anesthesiology. 1994 Nov;81(5):1149-61. doi: 10.1097/00000542-199411000-00008. PMID 7978473